CLINICAL TRIAL: NCT04235322
Title: Randomized, Placebo-controlled, Double-blind Study to Evaluate the Efficacy of 2LHERP® in Patients With Recurrent Genital Herpes Infections
Brief Title: Study of 2LHERP® in Genital Herpes Infections
Acronym: HEARTH-GEN
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Labo'life decided to end prematurely HEARTH-GEN study from April 18th 2023 due to very low recruitment rates (6/100). Labo'life decided to focus all its efforts on another study using 2LHERP® in herpes treatment, called HEARTH-OF (NCT04065971)
Sponsor: Labo'Life (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LLB-2019-01
Record Dates: First submitted 2020-01-16; First posted 2020-01-21 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Herpes Simplex, Genital
MeSH Terms: conditions — Herpes Genitalis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 2LHERP® arm (Experimental): 2LHERP® treatment (6 months of treatment)
  Interventions: Drug: 2LHERP®
- Placebo arm (Placebo Comparator): Placebo treatment (6 months of treatment)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 2LHERP® — The treatment schema consists in taking the content of one capsule a day, 15-30 minutes before breakfast, on an empty stomach, sequentially, according to capsules' numerical order: 1 through 10. When capsule number 10 is taken, capsule 1 of the next blister should be taken on the next day to continue the treatment. The duration of treatment will be 6 months of continuous intake of the content of 1 capsule/day.
  Other Names: 2LHERP
  Arms: 2LHERP® arm
Drug: Placebo — The treatment schema consists in taking the content of one capsule a day, 15-30 minutes before breakfast, on an empty stomach, sequentially, according to capsules' numerical order: 1 through 10. When capsule number 10 is taken, capsule 1 of the next blister should be taken on the next day to continue the treatment. The duration of treatment will be 6 months of continuous intake of the content of 1 capsule/day.
  Arms: Placebo arm

SUMMARY:
Herpes simplex virus (HSV) infection is very common, as most people will experience herpetic infection during their lifetime. The most common manifestation of HSV infection is sores which may appear at any age. No specific antiviral therapy is available to totally cure herpetic infections and today, there is no treatment that allows the definitive eradication of the virus.

The 2LHERP® has been available for more than 20 years, and has received a marketing authorization in Belgium by the FAMHP. It is used as an immune regulator in the treatment of herpetic infections. Since 2LHERP® has been made available, clinical observational data collected on treated patients have shown the beneficial effect on the disappearance of herpetic recurrences.

The purpose of this placebo-controlled trial is to evaluate the efficacy of 2LHERP® on the treatment of herpetic infections in adults.

DETAILED DESCRIPTION:
The study duration will be maximum 45 months with 33 months of inclusion and 12 months of follow-up. Patients aged between 18 and 80 years who present recurrent genital herpes infections (4 or more episodes within the 12-months' period prior to their study entry). The total number of patients to include will be 100 with 50 patients per group.

Primary objective:

Evaluation of the efficacy of 2LHERP® on the reduction of the number of recurrent genital herpes infections at 12 months compare to placebo.

Secondary objectives:

Comparison of the efficacy of 2LHERP® vs placebo, according to the following aspects:

* number of episodes at 6 months,
* remaining herpes infection recurrence free 6 and 12 months after the treatment initiation,
* time to first episode during the treatment,
* duration of episodes,
* symptomatology during the entire relapse time,
* use of Rescue Medication (RM),
* evaluation of impact on the quality of life,
* safety issues.

Treatment phase:

Group n°1 = 2LHERP® (6 months of treatment) Group n°2 = Placebo (6 months of treatment) Post-treatment follow-up phase: 6 months. Treatment will be considered successful if the number of herpetic episodes is reduced.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman aged 18-80 years,
* Patient presenting 4 or more episodes of genital herpes infections during the preceding 12-months' period (prior to the study entry),
* Woman of childbearing age under effective contraception,
* Patient reporting a current stable sexual relationship (steady sexual partner during study duration),
* Patient having faculties to understand and respect the constraints of the study,
* Signature of the Informed Consent Form.

Exclusion Criteria:

* Pregnant or breastfeeding woman,
* Patient under immunotherapy (including immunosuppressive treatment) or micro-immunotherapy received during last previous 6 months,
* Patient who had a suppressive antiviral therapy during last month,
* Patient who wishes to continue his/her suppressive antiviral therapy,
* Patient with known lactose intolerance,
* Patient who participated in a clinical study in the previous 3-month period,
* Patient who is not sufficiently motivated to engage in a follow-up period of 12 months, or likely to travel or to move before the end of the study,
* Patient with severe immunodeficiency disease requiring long term treatment (*) or under chemotherapy or radiotherapy or corticoid therapy,
* Patient under listed homeopathic or phytotherapy treatment,
* Patient using or addicted to recreational drugs.

(*) important renal or respiratory insufficiency, transplanted or grafted patients, HIV/AIDS, terminal cancer.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-01-25 (Actual); Primary Completion 2023-04-18 (Actual); Study Completion 2023-04-18 (Actual)

PRIMARY OUTCOMES:
Evaluation of the efficacy of 2LHERP® on the reduction of the number of recurrent genital herpes infections at 12 months compare to placebo. | 12 months
  Change from baseline within the number of episodes of genital herpes infection observed for 12 months, where the baseline value is the number of episodes experienced within the 12 months preceeding study enrolment.

SECONDARY OUTCOMES:
Comparison of the efficacy of 2LHERP® versus placebo according to the number of episodes at 6 months. | 6 months
  Number of episodes of herpes infections observed at month 6
Comparison of the efficacy of 2LHERP® versus placebo according to - remaining herpes infection recurrence free 6 and 12 months after the treatment initiation | 6 and 12 months
  Patient remaining herpes infection recurrence free 6 months and 12 months after the treatment initiation
Comparison of the efficacy of 2LHERP® versus placebo according to the time to first episode during the treatment | 6 months
  Time to first recurrence of herpes infection during the treatment
Comparison of the efficacy of 2LHERP® versus placebo according to the duration of episodes | 6 and 12 months
  Mean duration of episodes, the duration for a given episode being defined as the number of days between the start of the episode and the last day before all symptoms recorded as 'none' for 2 consecutive days, in the patient diary
Comparison of the efficacy of 2LHERP® versus placebo according to the symptomatology during the entire relapse time | 6 and 12 months
  Level of pain recorded daily on a visual analogue scale (100mm), as well as other associated symptomatology for genital (genital lesions/craks, difficulties to urinate, genital pruritus/burn, fever, QoL), which will be consequently measured as area under the curve (AUC)
Comparison of the efficacy of 2LHERP® versus placebo according to the use of Rescue Medication | 6 and 12 months
  Use of daily rescue medicine (RM), expressed with the cumulative number of days for the treatment period, the follow-up period and the entire study period
Comparison of the efficacy of 2LHERP® versus placebo according to the evaluation of impact on the quality of life | 6 and 12 months
  6-items questionnaire of quality of life
Comparison of the efficacy of 2LHERP® versus placebo according to safety issues | 6 months
  Adverse events (AEs) and severe adverse events (SAEs), considered as related or not to the study drug

CONTACTS AND LOCATIONS:
Locations (13):
- Belgium (13):
  - Private practice, Lodelinsart, Charleroi
  - Polyclinique D'Andenne, Andenne
  - Dr MANOUACH Fatiha, Brussels
  - Dr VERHEVEN Cécile, Brussels
  - Private Practice, Brussels
  - CHU Charleroi - Hopital Marie Curie, Charleroi
  - Cabinet privé, Gozée
  - Centre Hospitalier Regional de Huy, Huy
  - Private Practice, Libramont
  - Vivalia - Centre Hospitalier de L'Ardenne - Libramont Chevigny, Libramont
  - Dr PETTEAU Myriam, Nivelles
  - Dr ROULEFF Denis, Noirefontaine
  - Private Practice, Oisquercq

IPD SHARING:
Plan to Share IPD: No